CLINICAL TRIAL: NCT03866122
Title: Evaluating the Accuracy of a Neonatal Temperature Monitor in Comparison With Existing Temperature Monitors
Brief Title: Evaluation of a Novel Neonatal Temperature Monitor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: William Marsh Rice University (Other)
Collaborators: Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NTM-COMREC
Record Dates: First submitted 2019-01-03; First posted 2019-03-07 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Neonatal Hypothermia

STUDY DESIGN:
Intervention Model Description: One or more neonatal temperature monitors will be applied to the same infant; results between the monitors will be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neonatal Temperature Monitor (Experimental): One or more test devices (NTM, Bempu, Thermospot) will be attached to the infant in the neonatal intensive care unit (NICU) or KMC ward along with the Philips Intellivue patient monitor. Temperature will be monitored continuously using each device for up to 72 hours.
  Interventions: Device: NTM Monitoring

INTERVENTIONS:
Device: NTM Monitoring — NTM and a patient monitor will continuously collect temperature for up to 72 hours. Additionally, Bempu and Thermospot may monitor temperature for up to 72 hours.

SUMMARY:
A team of researchers at Rice University and Queen Elizabeth Central Hospital (QECH) are working to develop a low-cost temperature sensor that can continuously monitor an infant's temperature (NTM). This robust, low-cost device will allow for the individualized monitoring of each infant with alerts for hypo and hyperthermia. A reusable band placed around the infant's abdomen to hold the temperature sensor will eliminate disposable components. This study will assess the accuracy of this novel device against a gold standard (Philips Intellivue patient monitor) and up to two existing devices (Bempu and Thermospot).

DETAILED DESCRIPTION:
This study will assess the accuracy of this novel device against a commercially available patient monitor (Philips Intellivue MP30). Results will be compared to that of two existing devices designed for low resource settings: Bempu, a temperature monitor placed around an infant's wrist; and Thermospot, a sticker that changes color with temperature.

This study will enroll up to 150 infants at Queen Elizabeth Central Hospital. Up to 75 subjects will be collected from the neonatal ward and 75 subjects from the Kangaroo Mother Care (KMC) ward. This sample size will ensure that the investigators are able to collect sufficient data from infants with a range of gestational ages, weights, temperatures, and treatment locations (ie open cot, radiant warmer). The data from this study can be used to calculate the sample size needed in a larger study to evaluate changes in outcomes and nurse behavior related to the different temperature monitors (NTM, Bempu, Thermospot).

During the trial, the following steps will be taken:

A trained study nurse will assess the subject for clinical complications before attaching the temperature monitoring devices.

1. A trained study nurse or clinician will attach the test temperature monitoring devices to the infant. A trained research assistant from Rice University or from the Biomedical Engineering Department at Malawi Polytechnic will observe all procedures and will notify the nurse of any observed errors so they may be corrected. They will also be able to answer any technical questions from the nurse. If there is any concern for the comfort or skin of the infant, only one device may be placed on at a time (NTM, Bempu, ThermoSpot).
2. The trained study nurse will attach the temperature probe from the commercial gold standard as well as provide any other care needed.
3. A research assistant will use a laptop to collect data from the continuous temperature monitors (NTM and gold standard). The nurse will record the temperature readings every hour from all monitors on paper forms along with the standard of care.
4. Each time an alarm sounds from any device (Bempu and the commercial gold standard have audible alarms), the nurse will record all temperature values including a reading taken with the standard of care method. If the subject is found to be hyper/hypothermic, the nurse will respond with the appropriate standard of care.
5. Temperature monitoring will continue for up to 3 days. The research assistant may ask the nurse to remove and reapply the temperature probes during this period.

The goal of this study is to confirm the accuracy of these temperature monitors. Target accuracy for NTM device is +/- 0.5 C. In order to confirm this temperature accuracy in the settings of both the neonatal ward and the KMC ward, 75 subjects are needed in each setting. The international standards for clinical thermometers, standard number 80601-2-56, requires that 75 subjects from each patient population be tested to demonstrate the clinical accuracy of the thermometer. The clinical accuracy is reported using a measure of bias as well as the limits of agreement.

ELIGIBILITY:
Inclusion Criteria:

* The subject is currently being treated at QECH in the neonatal or KMC ward.
* Study devices are available for use.
* The subject's caregiver has provided informed consent for their child to participate.

Exclusion Criteria:

* At the clinician's discretion for any reason including, but not limited to:
* potential for skin irritation
* Cough
* other condition that may preclude use of the temperature belt
* concurrent treatments that may require increased patient care

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2022-09-06 (Estimated); Study Completion 2022-09-06 (Estimated)

PRIMARY OUTCOMES:
Temperature measurement accuracy | <72 hours
  Continuously measured temperature for test devices compared against Philips Intellivue patient monitor

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Richards-Kortum, PhD, Principal Investigator — William Marsh Rice University; Queen Dube, MD, Principal Investigator — Kamuzu University of Health Sciences
Locations (1):
- Rice University, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sosa Saenz SE, Hardy MK, Heenan M, Oden ZM, Richards-Kortum R, Dube Q, Kawaza K. Evaluation of a continuous neonatal temperature monitor for low-resource settings: a device feasibility pilot study. BMJ Paediatr Open. 2020 May 7;4(1):e000655. doi: 10.1136/bmjpo-2020-000655. eCollection 2020. PMID 32426530

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT03866122/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT03866122/ICF_001.pdf